CLINICAL TRIAL: NCT06284603
Title: The Effects of Hyperbaric Oxygen Therapy on Physical Capacity, Health, and Gut Microbiota in Healthy Male Adults
Brief Title: Effectiveness of Hyperbaric Oxygen Therapy in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWF_LA_HBOT
Record Dates: First submitted 2024-01-24; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: physical performance; vascular circulation; gut microbiota
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Two study groups (dependent on frequency of HBOT treatments) and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group 1: HBOT 3/week (Active Comparator): The protocol comprises 10 Hyperbaric Oxygen Treatments (HBOT), 3 sessions per week.
  Interventions: Device: Hyperbaric Oxygen Therapy - HBOT
- Study Group 2: HBOT 6/week (Active Comparator): The protocol comprises 10 Hyperbaric Oxygen Treatments (HBOT), 6 sessions per week.
  Interventions: Device: Hyperbaric Oxygen Therapy - HBOT
- Control Group (No Intervention): No changes to a daily routine.

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy - HBOT — Each session includes exposure of 60 minutes to 100% oxygen at 2.5 atmosphere absolute (ATA), with 5-minute air breaks every 20 minutes
  Arms: Study Group 1: HBOT 3/week; Study Group 2: HBOT 6/week

SUMMARY:
The goal of this controlled, experimental study is to learn about the effects of 10 sessions of hyperbaric oxygen therapy on physical performance, vascular circulation, biochemical parameters, and composition of the intestinal microbiota in young healthy men depending on the frequency of single treatments.

The main questions it aims to answer are:

1. Do 10 treatments of hyperbaric oxygen therapy induce significant changes in physical performance levels, vascular circulation, and concentrations of biochemical parameters in young, healthy men?
2. Does the body's response to 10 treatments of hyperbaric oxygen therapy differ depending on the frequency of treatments?
3. Does a series of hyperbaric oxygen therapy treatments induce significant changes in the composition of the intestinal microbiota, metabolome, and functional status of the intestines?

Participants are exposed to hyperoxia under hyperbaric conditions or form a control group with no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35;
* Healthy, physically active men;
* Subject who is knowingly willing to participate in the study;
* Subject able to read, understand and sign an informed consent to participate.

Exclusion Criteria:

* Inability to attend scheduled visits and/or follow study protocol;
* Use of HBOT prior to study inclusion;
* Severe or unstable physical impairment or severe cognitive deficits at study entry;
* Pressure-sensitive chest diseases (including moderate or severe asthma) or pressure-sensitive ear or sinus diseases;
* Active smoking;
* Having suffered an injury within 3 months up to the date of the study;
* Taking pre- and/or probiotics in the last 3 months before the study;
* Inpatient hospital or emergency room stay in the last 4 weeks prior to study entry;
* Travel to tropical countries during the last 4 weeks prior to the study;
* Taking antibiotics, steroids and steroid-anabolic agents during the last 4 weeks before the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Volume of oxygen and carbon dioxide | baseline and the next morning after the last HBOT intervention; up to 24 days.
  A cardiopulmonary exercise test (CPET) is conducted while an incremental running test on the treadmill using a portable breath-by-breath ergospirometer; VO2 and VCO2 are measured constantly.
Heart rate | baseline and the next morning after the last HBOT intervention; up to 24 days.
  Cardiopulmonary exercise test (CPET) is conducted while an incremental running test on the treadmill using a heart rate monitor.
Vascular circulation measures | baseline (before and immediately after CPET), before and after 5th treatment, and the next morning after the last HBOT intervention (before and immediately after CPET); up to 24 days.
  Nicotinamide adenine dinucleotide (NADH) content changes in the skin area are measured during transient ischemia and reperfusion with the use of the Flow Mediated Skin Fluorescence (FMSF) using The AngioExpert device (AngioExpert, Poland)

SECONDARY OUTCOMES:
Body composition (body mass, fat mass, lean body mass, muscle mass) | baseline and the next morning after the last HBOT intervention; up to 24 days.
  Body composition is tested by the dual X-ray absorptiometry method (DXA, Lunar Prodigy; General Electric Lunar Healthcare Technologies, Madison, USA).
Inflammatory cytokine profile | baseline and the next morning after the last HBOT intervention; up to 24 days.
  tumor necrosis factor (TNFalfa) and interleukins (IL-1beta, IL-6, IL-10) is measured using immunoenzymatic methods
Oxidative stress indicators | baseline and the next morning after the last HBOT intervention; up to 24 days.
  The activity of superoxide dismutase (SOD); catalase (CAT); glutathione peroxidase (GPx) is measured using spectrophotometric and immunoenzymatic methods
F2-Isoprostanes (F2-IsoP) | baseline and the next morning after the last HBOT intervention; up to 24 days.
  The measurement of F2-Isoprostanes (F2-IsoP) is performed using the spectrophotometric and immunoenzymatic methods
Brain-derived neurotrophic factor concentration (BDNF) | baseline and the next morning after the last HBOT intervention; up to 24 days.
  BDNF concentration is measured using immunoenzymatic methods
Nicotinamide (NAD) metabolites | baseline and the next morning after the last HBOT intervention; up to 24 days.
  NAD metabolites are measured using a combination of high-performance liquid chromatography-mass spectrometer methods (HPLC-MS)
Gut microbiome and metabolome | baseline and the next morning after the last HBOT intervention; up to 24 days.
  Metabolites produced by bacteria such as short-chain fatty acids (SCFA), tryptophan catabolites, and non-targeted metabolomes are measured using Ultra High Pressure Liquid Chromatography (UHPLC)
Indicators of intestinal inflammation (fecal calprotectin, claudin, occludin, zonulin, sIgA) | baseline and the next morning after the last HBOT intervention; up to 24 days.
  Indicators of intestinal inflammation are measured using Western blot analysis and real-time Polymerase Chain Reaction (RT-PCR).
endothelial nitric oxide synthase (eNOS) | baseline and the next morning after the last HBOT intervention; up to 24 days.
  eNOS activity is measured using immunoenzymatic methods
Vascular endothelial growth factor (VEGF) | baseline and after the intervention; up to 24 days.
  Concentration of VEGF is measured using immunoenzymatic methods
Hypoxia inducible factor-1 (HIF-1alfa) | baseline and the next morning after the last HBOT intervention; up to 24 days.
  Concentration of HIF-1alfa is measured using immunoenzymatic methods

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pospieszna, PhD., Principal Investigator — Department of Athletics, Strength and Conditioning, Poznan Univ of Physical Ed, Poznan, Poland
Locations (1):
- Poznan University of Physical Education, Poznan, Wielkopolska, Poland